CLINICAL TRIAL: NCT05245435
Title: Diagnostic and Prognostic Accuracy and Health Economics Considerations of [18F]-Fluoro-5α-dihydrotestosterone (FDHT)- Positron Emission Tomography (PET) and Circulating Tumor Cells - a Pilot Study in Patients Undergoing Cytoreductive Prostatectomy in the Setting of Primary Oligometastatic Prostate Cancer, in Patients With Primary Metastatic Hormone-sensitive Prostate Cancer, and in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Diagnostic and Prognostic Accuracy of FDHT-PET and Liquid Biopsies in Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was not possible with the chosen inclusion/exclusion criteria at our Institution.
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Zeitlinger, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FDHTProstate_Protocol_V3
Record Dates: First submitted 2021-09-28; First posted 2022-02-18 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- planned to undergo cytoreductive prostatectomy (Other): planned to undergo cytoreductive prostatectomy
  Interventions: Diagnostic Test: liquid biopsies
- newly diagnosed metastatic hormone-sensitive prostate cancer patients (Other): planned to undergo androgen deprivation therapy, and/or treatment with abiraterone acetate, and/or enzalutamide and/or docetaxel
  Interventions: Diagnostic Test: FDHT-PET Scan; Diagnostic Test: liquid biopsies
- metastatic castration-resistant prostate cancer patients (Other): who were not pre-treated with enzalutamide or abiraterone acetate and planned treatment with those drugs
  Interventions: Diagnostic Test: FDHT-PET Scan; Diagnostic Test: liquid biopsies
- primary oligometastatic hormone-sensitive prostate cancer patients (Other): who refuse to undergo cytoreductive radical prostatectomy will serve as control group
  Interventions: Diagnostic Test: liquid biopsies

INTERVENTIONS:
Diagnostic Test: FDHT-PET Scan — [18F]-fluoro-5α-dihydrotestosterone (FDHT)- positron emission tomography (PET)
  Arms: metastatic castration-resistant prostate cancer patients; newly diagnosed metastatic hormone-sensitive prostate cancer patients
Diagnostic Test: liquid biopsies — circulating tumor cell count and circulating tumor DNA abundance in blood of prostate cancer patients

SUMMARY:
Depending on the cohort of the study the diagnostic and prognostic accuracy and health economics considerations of [18F]-fluoro-5α-dihydrotestosterone (FDHT)- positron emission tomography (PET) and/or circulating tumor cells in prostate cancer patients are studied.

ELIGIBILITY:
Inclusion Criteria:

COHORT A:

* Age 18-75 years
* Histologically confirmed oligometastatic adenocarcinoma of the prostate (defined as ≤5 metastases in lymph node (LN) or bone)
* Eastern Cooperative Oncology Group (ECOG) Performance Status grade 0 or 1
* Planned cytoreductive radical prostatectomy
* ≤ 5 osseous and/or lymph node metastasis
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, questionnaire completion and other study procedures

COHORT B:

* Age 18-75 years
* Histologically confirmed oligometastatic adenocarcinoma of the prostate
* Newly diagnosed metastatic hormone-sensitive disease
* planned therapy with androgen deprivation therapy, and/or treatment with abiraterone acetate, and/or enzalutamide and/or docetaxel
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, questionnaire completion and other study procedures

COHORT C:

* Age 18-75 years
* Histologically confirmed oligometastatic adenocarcinoma of the prostate
* Metastatic castration-resistant disease
* Not pre-treated with enzalutamide or abiraterone acetate
* Planned therapy with abiraterone acetate, or enzalutamide
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, questionnaire completion and other study procedures

COHORT D (control group for Cohort A):

* Age 18-75 years
* Histologically confirmed oligometastatic adenocarcinoma of the prostate (defined as ≤5 metastases in lymph node (LN) or bone)
* Hormone-sensitive prostate cancer
* Refused cytoreductive radical prostatectomy
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, questionnaire completion and other study procedures

Exclusion Criteria:

COHORT A:

* HIV positive
* Any contraindication for surgery
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan
* Patient's not eligible for the size of the PET/MRI gantry

COHORTS B and C:

* HIV positive
* Any contraindication for tissue biopsy (if tissue biopsy is planned)
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan
* Patient's not eligible for the size of the PET/MRI gantry

COHORT D (control group for Cohort A):

* HIV positive
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan
* Patient's not eligible for the size of the PET/MRI gantry

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
FDHT total receptor expression (TRE) volume parameters compared to clinical follow-up | through study completion, an average of 2 years
FDHT total receptor expression (TRE) volume parameters compared to course of disease | through study completion, an average of 2 years
FDHT total receptor expression (TRE) volume parameters compared to androgen resistance | through study completion, an average of 2 years
FDHT total receptor expression (TRE) volume parameters compared to liquid biopsy parameters | through study completion, an average of 2 years
FDHT total receptor expression (TRE) volume parameters compared to IHC patterns | through study completion, an average of 2 years
FDHT total receptor expression (TRE) volume parameters compared to stage of disease | through study completion, an average of 2 years
CTC count before and after treatment | through study completion, an average of 2 years
ctDNA abundance before and after treatment | through study completion, an average of 2 years
(Quantitative) IHC analysis of androgen specific receptor expression levels (FDHT) in tissue | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No